CLINICAL TRIAL: NCT03170700
Title: Use of Engaging Online Videos in Conjunction With New Feeding Content to Enhance a Current EFNEP Program in the Prevention of Child Obesity
Brief Title: Online Videos and New Feeding Content to Enhance a Current EFNEP Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Washington State University (Other); Colorado State University (Other)
Responsible Party: Principal Investigator, Sheryl Hughes, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-36455; 2015-68001-23311 (Other: USDA)
Record Dates: First submitted 2017-05-08; First posted 2017-05-31 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Childhood
Keywords: preschool; eating behaviors; family
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: 1) Nutrition Program (Eating Smart • Being Active) alone (control); 2) Nutrition program with parental feeding content (In-person); or 3) Nutrition program with parental feeding content (online).
Who Masked: Outcomes Assessor
Masking Description: Assessments will be conducted by staff blind to group membership.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will receive a nutrition program without parental feeding content. They will attend the nutrition program (Eating Smart • Being Active).
- In-person (Experimental): Nutrition program with in-person parental feeding content.
  Interventions: Behavioral: Nutrition program with in-person parental feeding content
- Online (Experimental): Nutrition program with online parental feeding content.
  Interventions: Behavioral: Nutrition program with online parental feeding content

INTERVENTIONS:
Behavioral: Nutrition program with in-person parental feeding content — Participants will attend the nutrition program (Eating Smart • Being Active) and be provided with in-person parental feeding content.
  Arms: In-person
Behavioral: Nutrition program with online parental feeding content — Participants will attend the nutrition program (Eating Smart • Being Active). They will access parental feeding content online.
  Arms: Online

SUMMARY:
The goal of this study is to further increase the impact of a validated and widely-used Eating Smart • Being Active EFNEP curriculum by teaching parents responsive feeding practices resulting in the development of healthier patterns of child eating behavior and food intake. Additionally, the effectiveness of two delivery strategies for adding feeding video-based content will be examined (in-person versus online lessons).

DETAILED DESCRIPTION:
During Phase I of the project (first two years), the leadership team composed of both research and extension investigators will work with the media production team to edit the SEEDS videotapes to meet the needs of the current project and to develop the website and activities for use in the online condition. Phase II (second three years) will be a large scale evaluation of this program. In this phase, classes of EFNEP participants in Colorado and Washington will be randomly assigned to one of three conditions: 1) Eating Smart • Being Active alone (control); 2) Eating Smart • Being Active plus feeding videos at the weekly EFNEP sessions, plus facilitated group discussion (in-person); or 3) Eating Smart • Being Active plus online videos and activities, (online). Pre- and post-program assessments, 6- and 12-month follow ups will be conducted to assess responsive feeding, providing structure, food exploration, child eating behaviors, parent knowledge, and child dietary intake. Child dietary intake will be obtained on a sub-sample of 90 participants. In Phase III, the investigators will begin dissemination.

A total of 543 participants were recruited in five locations to participate in the project: 262 from three counties in Colorado and 281 from three counties in Washington (English and Spanish participants). A total of 4 to 10 mothers were recruited for each group. After recruitment, groups were randomly assigned to the three conditions ensuring a relatively equal number of participants per condition.

Data from children who have any kind of food allergies or diabetes or are on special diet will be excluded from the analyses.

To ensure program fidelity, program educators will complete implementation checklists, and 20% of the sessions will be attended by an additional grant staff member to conduct implementation observations and assess participant engagement. Detailed records of participant attendance will be collected to assess dosage effects and attrition. All assessments will be conducted by grant project staff blind to the group status of the participants. Retention of participants will be maximized using strategies such as obtaining multiple phone numbers for each family; obtaining external contact information for siblings and close friends; sending interim reminders with the goal of fostering contact should the family move; and phone calls, emails or letters between data collection points to each family.

ELIGIBILITY:
Inclusion Criteria:

* Parents who attend EFNEP programs in the states of WA and CO.

Exclusion Criteria:

* Parents with children younger than age 2 and older than age 8 will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Responsive Feeding from the modified Child Feeding Questionnaire | Up to 12-month follow up
  Five subscales measuring responsiveness, restriction, use of food as reward, monitoring, and pressure to eat will be assessed using a 5-point Likert scale. Parents will report on these constructs that assess responsive feeding.
Providing Structure from the modified Child Feeding Questionnaire | Up to 12-month follow up
  Seven subscales measuring parent decides on portions, family meals, serves measured portions, child helps prepare, eat whenever, indulgent feeding, and eat at regular times will be assessed using a 5-point Likert scale. Parents will report on these constructs that assess responsive feeding.
Novel Foods from the modified Child Feeding Questionnaire | Up to 12-month follow up
  Four subscales measuring encouraging exploration, offering new foods, urging new foods, and low pressure strategies for encouragement will be assessed using a 5-point Likert scale. Parents will report on these constructs that assess responsive feeding.

SECONDARY OUTCOMES:
Parental Knowledge Questionnaire | Up to 12-month follow up
  A questionnaire measuring aspects of feeding and nutrition knowledge and content covered in the prevention curriculum will be assessed.
Child Eating Behaviors | Up to 12-month follow up
  Parental report of child eating behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O Hughes, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Washington State University, Pullman, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Power TG, Baker SS, Barale KV, Aragon MC, Lanigan JD, Parker L, Garcia KS, Auld G, Micheli N, Hughes SO. Using Mobile Technology for Family-Based Prevention in Families with Low Incomes: Lessons from a Randomized Controlled Trial of a Childhood Obesity Prevention Program. Prev Sci. 2024 Feb;25(2):369-379. doi: 10.1007/s11121-023-01637-8. Epub 2024 Feb 7. PMID 38321316
- [Derived] Hughes SO, Power TG, Baker SS, Barale KV, Aragon MC, Lanigan JD, Parker L, Silva Garcia K, Auld G, Johnston CA, Micheli N. Short-Term Efficacy of a Childhood Obesity Prevention Program Designed to Pair Feeding Content With Nutrition Education. Child Obes. 2023 Jun;19(4):239-248. doi: 10.1089/chi.2022.0030. Epub 2022 Jun 16. PMID 35708621